CLINICAL TRIAL: NCT06750562
Title: The Effect of Interactive Game Supported Sleep Hygiene Training on Sleep Quality, Menopausal Symptoms and Quality of Life in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meryem Vural Şahin (Other)
Responsible Party: Sponsor-Investigator, Meryem Vural Şahin, PHD Student, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 913715751
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Menopause; Sleep

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental intervention (Experimental): This group will receive online sleep hygiene training for 4 weeks. The training will be given one day a week and last 30 minutes.
  is foreseen. After each training, an interactive sleep hygiene game will be shared online. A total of 4 interactive sleep hygiene games will be shared. The total duration of a game will not exceed 20 minutes.
  Interventions: Behavioral: interactive game
- control group (No Intervention): this group will be given online sleep hygiene training once a week for a total of 4 weeks. The duration of each training will not exceed 30 minutes.

INTERVENTIONS:
Behavioral: interactive game — Interactive game supported sleep hygiene will be prepared by researchers. The game will be shared after each sleep hygiene training. The intervention is planned as 4 trainings and 4 games in total.
  Arms: experimental intervention

SUMMARY:
This study will present an innovative approach for sleep hygiene education in this age group by developing an interactive game-based education model for menopausal women. Gamification methods enable education to be made more interactive, engaging and fun, which can improve the learning process. Considering the lack of such an application in the literature, this study is thought to fill a gap both in Turkey and worldwide. While health education is usually presented with classical methods, interactive gamification methods have attracted more attention in recent years. This study is thought to be one of the first to show how gamification can be used in menopausal women. In addition, the findings of the study may show that improving sleep hygiene in the menopausal period may provide positive effects not only on sleep quality, but also on menopausal symptoms and overall quality of life. Therefore, it is thought that the study may provide critical data in both symptom management and women's health. It is thought that this study will pioneer the development of new education and counselling models in the field of midwifery. Especially midwives can take a more effective role in symptom management by using such interactive trainings for women in menopausal period. Thus, it is thought that an innovative approach will be brought to midwifery education and practices.

DETAILED DESCRIPTION:
Sleep hygiene training requires the acquisition and practice of specific behaviours, but is typically delivered in a single meeting with a practitioner. Such formats may not encourage participation or provide opportunities to review and practice behaviours. An alternative format, game-based learning, provides interaction with activities that have a clear set of objectives, constraints and rules. The digital game creates an individual communication environment that incorporates the digitality, interactivity, virtuality, variability, modularity features of the new communication environment and incorporates these features into the act of playing games. Compared to traditional education, game-based education provides situated learning as it can mimic the real world in which the learner is situated. In educational research, it is emphasised that the game factor increases motivation. In a meta-analysis of 22 studies on video game-based interventions targeting healthy adults older than 44 years, it was found that video game-based interventions had positive effects on objectively measured physical and social health.

Midwives play a critical role in meeting basic human needs and supporting the independence of individuals. One of the most basic needs of menopausal women is the need for sleep. However, in the national and international literature, there is no interactive game-supported web-based sleep hygiene training application for menopausal women. This situation reveals the need to develop an innovative approach in which midwives can provide more effective education and counselling in symptom management. Interactive game-based education was planned to provide a new and effective method to support women's health by increasing knowledge about sleep hygiene in menopausal women and to strengthen the role of midwives in this process.

ELIGIBILITY:
Inclusion Criteria:

* Score >5 according to the PDCI
* No problem in speaking and understanding Turkish
* Being in the menopausal period between the ages of 40-60
* Not having a systemic disease (rheumatoid arthritis, multiple sclerosis, etc.).
* Volunteering to participate in the study
* Absence of menstruation in the last 12 months
* Natural menopause
* Not working in a shift job
* Having the appropriate devices to play the game (computer, smartphone and internet connection)

Exclusion Criteria:

* - Receiving Hormone Replacement Therapy
* Diagnosed psychiatric illness
* Receiving a cancer diagnosis
* Entering menopause for surgical reasons
* Presence of chronic pain
* Diagnosis of a sleep disorder
* Receiving pharmacological or nonpharmacological treatment for sleep disorder

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — in menopause
Enrollment: 82 (Actual)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-09-27 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 1 month after the training and interactive game application
  The total score varies between 0-21. A total score higher than 5 indicates 'poor sleep quality'.
Menopause Symptoms Assessment Scale (MSAS) | 1 month after the training and interactive game
  The lowest score of 0 (zero) and the highest score of 44 (forty-four) can be obtained from the MSAS. The increase in the total number of points of the scale reveals an increase in the severity of menopausal symptoms in women experiencing menopausal symptoms.
Menopause Specific Quality of Life Scale (MSQOL) | 1 month after the training and interactive game application
  The lowest score that can be obtained from the total scale is '0' and the highest score (29X6) is 154.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gülhane Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seaver C, Bowers C, Beidel D, Holt L, Ramakrishnan S. A game-based learning approach to sleep hygiene education: a pilot investigation. Front Digit Health. 2024 Apr 12;6:1334840. doi: 10.3389/fdgth.2024.1334840. eCollection 2024. PMID 38680214
- [Background] Vazquez FL, Otero P, Garcia-Casal JA, Blanco V, Torres AJ, Arrojo M. Efficacy of video game-based interventions for active aging. A systematic literature review and meta-analysis. PLoS One. 2018 Dec 11;13(12):e0208192. doi: 10.1371/journal.pone.0208192. eCollection 2018. PMID 30533015
- [Background] Chung KF, Lee CT, Yeung WF, Chan MS, Chung EW, Lin WL. Sleep hygiene education as a treatment of insomnia: a systematic review and meta-analysis. Fam Pract. 2018 Jul 23;35(4):365-375. doi: 10.1093/fampra/cmx122. PMID 29194467
- [Background] Kalmbach DA, Cheng P, Arnedt JT, Cuamatzi-Castelan A, Atkinson RL, Fellman-Couture C, Roehrs T, Drake CL. Improving Daytime Functioning, Work Performance, and Quality of Life in Postmenopausal Women With Insomnia: Comparing Cognitive Behavioral Therapy for Insomnia, Sleep Restriction Therapy, and Sleep Hygiene Education. J Clin Sleep Med. 2019 Jul 15;15(7):999-1010. doi: 10.5664/jcsm.7882. PMID 31383238
- [Background] Abdelaziz EM, Elsharkawy NB, Mohamed SM. The relationship between sleep quality and menopausal symptoms among postmenopausal women in Saudi Arabia. Saudi Med J. 2022 Apr;43(4):401-407. doi: 10.15537/smj.2022.43.4.20210682. PMID 35414619
- [Background] Johnson A, Roberts L, Elkins G. Complementary and Alternative Medicine for Menopause. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X19829380. doi: 10.1177/2515690X19829380. PMID 30868921
- [Background] Schaedel Z, Holloway D, Bruce D, Rymer J. Management of sleep disorders in the menopausal transition. Post Reprod Health. 2021 Dec;27(4):209-214. doi: 10.1177/20533691211039151. Epub 2021 Nov 8. PMID 34748453
- [Background] Song Z, Jiang R, Li C, Jin F, Tao M. Menopausal Symptoms and Sleep Quality in Women Aged 40-65 Years. Biomed Res Int. 2022 Aug 9;2022:2560053. doi: 10.1155/2022/2560053. eCollection 2022. PMID 35983252
- [Background] Tandon VR, Sharma S, Mahajan A, Mahajan A, Tandon A. Menopause and Sleep Disorders. J Midlife Health. 2022 Jan-Mar;13(1):26-33. doi: 10.4103/jmh.jmh_18_22. Epub 2022 May 2. PMID 35707298
- [Background] Lucena L, Santos-Junior JG, Tufik S, Hachul H. Effect of a lavender essential oil and sleep hygiene protocol on insomnia in postmenopausal women: A pilot randomized clinical trial. Explore (NY). 2024 Jan-Feb;20(1):116-125. doi: 10.1016/j.explore.2023.07.004. Epub 2023 Jul 17. PMID 37495431
- [Background] Ha B, Kim J, So WY, Kim S. Effects of Nonpharmacological Interventions on Sleep Quality and Insomnia in Perimenopausal and Postmenopausal Women: A Meta-Analysis. Healthcare (Basel). 2023 Jan 22;11(3):327. doi: 10.3390/healthcare11030327. PMID 36766902